CLINICAL TRIAL: NCT06732102
Title: PhillyCEAL: Addressing Disparities in Chronic Disease Self-management Through an Enhanced Community Health Worker Program
Brief Title: Philly CEAL- DECIDE+ Adaptation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Westat (Other); City of Phladelphia - Office of Community Empowerment and Opportunity (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 856216
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Disparities; Community Health Workers; Cardiovascular Diseases; Social Determinants of Health (SDOH)
Keywords: Community Health Worker; Chronic Disease Management; Cardiovascular Health; Unmet social needs
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants can choose whether they wish to participate in the DECIDE group sessions or engage in traditional CHW services, yet they will be randomized to receive either one or two calls per month from their designated community health worker. A 1:1 randomization process will be employed, whereby each individual is assigned a random number generated by a computer algorithm. Participants with an even number will be allocated to receive one call per month (the current standard of care), while those assigned an odd number will receive two calls per month. This random assignment ensures an equal probability of assignment to each group, minimizing selection bias and supporting balanced distribution across the study conditions participation in the DECIDE intervention vs no DECIDE sessions. Participants will be blinded to their assigned call schedule and will be notified at the end of the trial as part of the dissemination of study results.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DECIDE+ Arm with Biweekly Follow-up Calls (Experimental): We will offer the DECIDE intervention as a group-based program. This program, facilitated by CHWs, will emphasize the importance of observational learning and group support to strengthen their CVD problem solving. Consistent with the DECIDE intervention's existing evidence-base, CVD problem solving is hypothesized to strengthen an individual's CVD self-management self-efficacy and skills, respectively. Increased self-management self-efficacy and skills are posited to increase the adoption of CVD-related health promotive behaviors. Participants in this arm will also receive 2 follow-up calls per month from their assigned CHW.
  Interventions: Behavioral: DECIDE; Behavioral: Community Health Worker Support
- DECIDE+ Arm with a Monthly Follow-up Call (Experimental): We will offer the DECIDE intervention as a group-based program. This program, facilitated by CHWs, will emphasize the importance of observational learning and group support to strengthen their CVD problem solving. Consistent with the DECIDE intervention's existing evidence-base, CVD problem solving is hypothesized to strengthen an individual's CVD self-management self-efficacy and skills, respectively. Increased self-management self-efficacy and skills are posited to increase the adoption of CVD-related health promotive behaviors. Participants in this arm will also receive 1 follow-up call per month from their assigned CHW.
  Interventions: Behavioral: DECIDE; Behavioral: Community Health Worker Support
- CHW Standard of Care with Biweekly Follow-up Calls (Active Comparator): CHWs currently serve Philadelphia residents by offering a wide range of personalized services aimed at improving their well-being. CHWs act as a crucial link between communities and healthcare providers, helping residents navigate the healthcare system. By offering guidance and social assistance, they improve community members' ability to communicate effectively with healthcare professionals. They also deliver health education that is culturally and linguistically appropriate, advocate for the health of individuals and communities, coordinate care through referrals and follow-up services, and assist eligible individuals in enrolling in federal, state, local, or nonprofit health and human services programs. Participants in this arm will receive a biweekly CHW Follow-up call.
  Interventions: Behavioral: Community Health Worker Support
- CHW Standard of Care with Monthy Follow-up Calls (Active Comparator): CHWs currently serve Philadelphia residents by offering a wide range of personalized services aimed at improving their well-being. CHWs act as a crucial link between communities and healthcare providers, helping residents navigate the healthcare system. By offering guidance and social assistance, they improve community members' ability to communicate effectively with healthcare professionals. They also deliver health education that is culturally and linguistically appropriate, advocate for the health of individuals and communities, coordinate care through referrals and follow-up services, and assist eligible individuals in enrolling in federal, state, local, or nonprofit health and human services programs. Participants in this arm will receive a Monthly CHW Follow-up call.
  Interventions: Behavioral: Community Health Worker Support

INTERVENTIONS:
Behavioral: DECIDE — Decision-making Education for Choices In Diabetes Everyday (DECIDE) is a self-management program in which education and problem-solving training are utilized to promote behavior change for optimal clinical outcomes.
  Arms: DECIDE+ Arm with Biweekly Follow-up Calls; DECIDE+ Arm with a Monthly Follow-up Call
Behavioral: Community Health Worker Support — CHWs are expected to actively equip individuals and communities by enhancing health knowledge and promoting self-sufficiency through various activities such as outreach, community education, informal counseling, social support, and advocacy. They act as a crucial link between communities and healthcare providers, helping residents navigate the healthcare system. By offering guidance and social assistance, they improve community members' ability to communicate effectively with healthcare professionals. They also deliver health education that is culturally and linguistically appropriate, advocate for the health of individuals and communities, coordinate care through referrals and follow-up services, and assist eligible individuals in enrolling in federal, state, local, or nonprofit health and human services programs.

SUMMARY:
Cardiovascular disease (CVD) disproportionately affects racial/ethnic minorities and underserved populations in Philadelphia. This study aims to evaluate the effectiveness of an enhanced community health worker (CHW) program that combines the evidence-based DECIDE self-management intervention with structured CHW consultations to improve CVD self-management skills and address social needs. Using a Type 1 Hybrid Effectiveness-Implementation Design, we will recruit 500 Philadelphia residents aged 35-75 with CVD risk factors and unmet social needs. Participants will be offered the DECIDE+ intervention (9 bi-weekly group sessions plus alternating CHW consultations) or continue with standard CHW services. The primary outcome is CVD self-management skills measured by the Self-care of Chronic Illness Inventory Maintenance scale. Secondary outcomes include health behaviors and resolution of social needs. Implementation outcomes will assess CHW experiences, community advisory council impact, and factors influencing participation. Propensity score methods will be used to compare changes in outcomes between DECIDE+ participants and those receiving standard CHW services. Mediation analyses will examine pathways through problem-solving skills, self-efficacy, and social needs resolution. Mixed methods will evaluate implementation outcomes. This study will provide evidence on the effectiveness of integrating an evidence-based self-management program with CHW services to address both clinical and social needs.

This study has the potential to generate important and impactful findings that can advance health equity and the science of effective community health worker programs. By rigorously evaluating the real-world implementation of a city-wide CHW-delivered chronic disease self-management program that also addresses collaborative approaches and support to addressing social needs, our findings can provide a roadmap for other communities looking to implement evidence-based interventions to reduce health disparities. Demonstrating improved CVD self-management behaviors and reduced social needs among Philadelphia residents receiving the DECIDE+ intervention would provide compelling evidence for the synergistic benefit of these services, and to sustain and scale up this model.

OBJECTIVES: We propose both effectiveness and implementation questions to guide our work:

Effectiveness of CHW Engagement:

1. Is the DECIDE intervention with CHW consultations (DECIDE+) effective in improving CVD self-management skills compared to the standard and limited CHW engagement?

   1. Do DECIDE+ sessions improve CVD self-management skills by strengthening problem solving and self-efficacy?
   2. Does participation in CHW consultations improve CVD self-management skills by meeting social needs?

   Implementation Questions:
2. What key sociodemographic and psychosocial factors influence client participation in the study?
3. How do CHWs perceive the impact of facilitator training on their a.) knowledge, attitudes and practices in supporting clients b.) personal health management, and c.) job satisfaction?
4. How does the CAC facilitate resource mobilization to enhance access to services that address social needs in Philadelphia's communities?

DETAILED DESCRIPTION:
The American Heart Association estimates that a person dies every 33 seconds from cardiovascular disease (CVD). CVD remains a leading cause of mortality in the US. Even people with just one risk factor for CVD (e.g. hypertension) have an estimated 30% lifetime risk of experiencing a cardiovascular event (e.g. heart attack); this risk increases to 70% among people with 2 or more risk factors. Therefore, there remains an urgent need to improve cardiovascular health behaviors and decrease risk for CVD particularly among racial/ethnic minoritized populations who are disproportionately affected by CVD and associated risk factors. Compared to Non-Latino Whites, Blacks experience higher rates of CVD risk factors - particularly obesity and hypertension - and are more likely to die from CVD. Similarly, higher prevalence and mortality of ischemic heart disease are noted in some Asian-American subgroups when compared to non-Latino Whites. Although, Latinos do not experience higher rates of CVD mortality compared to non-Latino Whites, Latinos are experiencing increasing rates of stroke and heart-failure related mortality. For those with CVD risk factors such as hypertension, diabetes, and hyperlipidemia, optimal management of these conditions can improve quality of life and reduce risk for premature mortality. Despite bordering the healthiest county in Pennsylvania, Philadelphia is the least healthy county in Pennsylvania and one of the least healthy in the nation. Compared to higher ranked counties in Pennsylvania, Philadelphians report less cardiovascular health behaviors (e.g. less physical activity, more smoking).

Chronic disease self-management (CDSM) is an evidence-based approach for chronic disease control, reducing health care utilization, and improving quality of life at the individual level. CDSM refers to a set of ongoing processes to proactively manage one's health condition(s). These processes can be categorized as - 1) disease/condition specific knowledge, 2) self-regulation skills including problem-solving, action planning, and effective coping, and 3) engaging social support. DECIDE (Decision-making Education for Choices in Diabetes Everyday) is a 9-session self-management program delivered bi-weekly for 90-minutes that offers disease specific education and problem-solving training for behavior change and optimal chronic disease management. DECIDE was originally developed for African Americans with diabetes and low-literacy, and has been modified for other populations and for other cardiovascular conditions including hypertension, heart failure, and chronic kidney disease. However, for programs like DECIDE to be effective they must be accessible to the target population, and people need supportive environments (e.g. stable housing) to realize optimal chronic disease management.

Community health workers (CHWs) are an essential community-level resource for the implementation and sustainability of self-management programs for under-resourced, racial/ethnic minoritized populations. For many underserved populations, SDoH inequities (e.g. neighborhood deprivation, access to health insurance) impede consistent CDSM. SDoH are determined by macro-level factors (e.g. organizational and civic systems and policies) that influence individual level social needs such as food and housing security. A key element of CHW effectiveness for promoting self-management among community members is their ability to provide ongoing support and advocacy for navigating the complex social determinants of health to address individual social needs. There is compelling evidence demonstrating the benefit and cost-effectiveness of CHW services for promoting CDSM and improving health outcome. Specifically in Philadelphia, CHW support for addressing social needs and helping with health system navigation has reduced all cause hospitalization and hospital stay among a low-income and high-risk for CVD population.

Recognizing the reciprocal determinism between individuals, their environment, and their behaviors, our DECIDE+ intervention integrates components to enhance CVD self-management. At the individual level, we will offer the DECIDE intervention as a group-based program. This program, facilitated by CHWs, will emphasize the importance of observational learning and group support to strengthen their CVD problem solving. Consistent with the DECIDE intervention's existing evidence-base, CVD problem solving is hypothesized to strengthen an individual's CVD self-management self-efficacy and skills, respectively. Increased self-management self-efficacy and skills are posited to increase the adoption of CVD-related health promotive behaviors.

At the community level, we also recognize that individuals' social environment may deter individuals' willingness and/or ability to engage in CVD-related health promotive behaviors if they have more pressing social needs requiring attention. Therefore, we propose to supplement the DECIDE intervention with biweekly one on one consultations with CHWs to address their environmental and situational barriers. By offering continued engagement with CHWs, we expect that participants will have greater success in meeting their social needs. As noted above, our CAC will support these efforts by identifying solutions and leveraging community resources that may further address participants' environmental and situational barriers. Ultimately, we posit that participants who have their social needs met will be more likely to engage in CVD-related self-management skills and health promotive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Philadelphia
* Be between 35 and 75 years of age (inclusive)
* Self-report having been told by a healthcare provider that they have one or more of the following CVD-related chronic conditions:

  1. Pre-diabetes
  2. Diabetes
  3. Hypertension
  4. Hyperlipidemia/ high cholesterol)
  5. BMI >=30.
* Have completed an initial visit with a CEO CHW
* Have one or more unmet social needs identified in the CEO Intake Form in the following areas:

  1. Housing Stability,
  2. Food security,
  3. Transportation to medical appointments and/or work,
  4. Employment,
  5. Household utilities,
  6. Healthcare access,
  7. Health literacy, and
  8. Social support.
* Willing to consent to participate in the CEAL study regular access to a mobile device to qualify for enrollment.

Exclusion Criteria:

* Does not reside in Philadelphia
* Not between 35 and 75 years of age (inclusive)
* Does not self-report having been told by a healthcare provider that they have one or more of the following CVD-related chronic conditions:

  1. Pre-diabetes
  2. Diabetes
  3. Hypertension
  4. Hyperlipidemia/ high cholesterol)
  5. BMI >=30.
* Has not completed an initial visit with a CEO CHW
* Does not have one or more unmet social needs identified in the CEO Intake Form in the following areas:

  1. Housing Stability,
  2. Food security,
  3. Transportation to medical appointments and/or work, employment,
  4. Household utilities,
  5. Healthcare access,
  6. Health literacy, and
  7. Social support.
* Unwilling to consent to participate in the CEAL study regular access to a mobile device to qualify for enrollment.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
CVD Self-Management Skills | From enrollment to the end of follow-up period at 6 months
  CVD self-management skills, measured by the Self-care of Chronic Illness Inventory Maintenance scale (SC-CII Maintenance).(Riegel et al., 2018) This 8-item measure of self-care maintenance assesses the degree to which an individual with chronic illness uses various strategies to maintain physical and emotional stability and includes both health promoting behaviors and illness-related behaviors. The scale is scored by summing the responses on the eight items and dividing by the total possible points to create a scale ranging from 0-1, where higher scores indicate better self-care maintenance.

SECONDARY OUTCOMES:
Unmet Social Needs | From enrollment to the end of follow-up at 6 months
  We will also assess participants' unmet social needs and their appropriate resolution, as measured using an 8-domain social needs inventory. For each social need identified, the degree to which the need has been addressed by a CHW will be assessed by asking participants whether they have discussed this need with a CHW, whether they have received a referral for this need form their CHW, and whether they have followed up on that referral. These follow up questions will be used to create a continuum score ranging from 0-3 for each social need, and a total social needs resolution score will be calculated by dividing the sum of the participants score across identified needs by the total possible score given the number of needs identified to create a scale ranging from 0-1, where higher scores indicate greater resolution of social needs.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bauermeister, MPH, PhD, Principal Investigator — University of Pennsylvania; Antonia Villarruel, RN, PhD, Principal Investigator — University of Pennsylvania; Carmen Alvarez, RN, PhD, Principal Investigator — University of Pennsylvania; Stephen Bonett, RN, PhD, Principal Investigator — University of Pennsylvania; Ashley Clemmons, Principal Investigator — Office of Community Empowerment and Opportunity
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will gather information from at least 500 Philadelphia residents, most of whom will be ethnic/minorities. We will gather IPD via survey domains included in Common Survey 4 (e.g., sociodemographic characteristics, health status, health behaviors). We will also ask participants questions about their satisfaction with the DECIDE intervention, and experiences with Community Health Workers. De-identified data for this project will be deposited into the NIH CEAL Repository. The data and documentation will undergo a mandatory review by WESTAT data curators to ensure that they are accessible, organized, and well documented. We will make updates to our dataset according to the suggestions of the data curators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months and ending 3 years after the publication of results.
Access Criteria: Data will be findable through the CEAL Repository database that has been established. The study will be assigned a digital object identifier (DOI). We will assure the timely release and sharing of data no later than the acceptance for publication of the main findings from the final dataset and will protect the rights and privacy of human subjects who participate in sponsored research by redacting all identifiers, and adopting other strategies to minimize risks of unauthorized disclosure of personal identifiers.
URL: https://www.nihceal.org/

REFERENCES:
- See also: Study Website — http://www.phillyceal.org